CLINICAL TRIAL: NCT05377567
Title: Cost-utility and Immuno-inflammatory Underpinnings of the FIBROWALK Multicomponent Therapy in Online or Outdoor Format in Fibromyalgia: a Randomised, Controlled Trial (the On&Out Study)
Brief Title: Cost-utility and Immuno-inflammatory Effects of the FIBROWALK in Patients With Fibromyalgia (the On&Out Study)
Acronym: On&Out
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Universitat Autonoma de Barcelona (Other); Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ON&OUT
Record Dates: First submitted 2022-05-04; First posted 2022-05-17 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; Cost-utility; multicomponent treatment; randomized controlled trial; Biomarkers
MeSH Terms: conditions — Fibromyalgia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAU + FIBRO-On (Experimental): FIBRO-On is a virtual multicomponent non-pharmacological program based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness Training
  Interventions: Behavioral: TAU + FIBRO-On
- TAU + FIBRO-Out (Active Comparator): FIBRO-Out is a outdoor multicomponent non-pharmacological program based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness Training
  Interventions: Behavioral: TAU + FIBRO-Out
- Treatment as Usual (TAU) (Active Comparator): Treatment-as-Usual (TAU) consisted of the prescribed drugs adapted to the symptomatic profile of each patient and basic face to face and written advice on PNE and aerobic exercise adapted to the physical capacities of the patients at the beginning of the study.patient
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: TAU + FIBRO-On — Group treatment protocol of 12 weekly 60 minute sessions (virtual intervention)
  Arms: TAU + FIBRO-On
Behavioral: TAU + FIBRO-Out — Group treatment protocol of 12 weekly 120 minute sessions (outdoor intervention)
  Arms: TAU + FIBRO-Out
Other: Treatment as Usual (TAU) — Standard pharmacological treatment usually provided to patients with fibromyalgia.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The present project will evaluate through a randomised controlled clinical trial with 6-month follow-up, the efficacy and cost-utility (6-month time horizon) of the multicomponent FIBROWALK programme in an online (i.e., FIBRO-On) and outdoor (i.e., FIBRO-Out) adjunctive to usual care (HC) format, as compared to HC. In order to determine the mechanisms of action of the clinical effects of the interventions studied 6 months after the start of treatment, pre-post changes will be evaluated in various psychological variables considered to be mediators from a theoretical point of view, as well as in immuno-inflammatory markers with evidence of alteration in FM and/or potentially modifiable by the interventions proposed (i.e. IL-6, CXCL8, IL-17A, IL-4, IL-10, high-sensitivity C-reactive protein). In the field of personalised treatment in chronic pain, the design of the present study with 3 treatment branches will also make it possible to establish whether certain patient profiles or baseline psychobiological characteristics can predict the short- and medium-term clinical response to the treatments studied.

DETAILED DESCRIPTION:
Introduction: The On&Out study is aimed at assessing the efficacy, cost-utility and immuno-inflammatory underpinnings of the FIBROWALK multicomponent intervention conducted in two different settings: online (FIBRO-On) or outdoors (FIBRO-Out). Both interventions have proved to be efficacious in the short-term but there is no study assessing their comparative efficacy nor their long-term effects. This study will also evaluate the cost-utility (6-month time-horizon) and the effects in blood biomarkers level of both interventions for the first time. The objectives of this 6-month, randomized, controlled trial (RCT) are (i) to examine the efficacy and cost-utility of adding FIBRO-On or FIBRO-Out to treatment-as-usual (TAU) for individuals with fibromyalgia; (ii) to identify pre-post differences in levels in blood biomarkers in the three study arms and (iii) to analyze the role of some psychological process variables as mediators of 6-month clinical outcomes. Methods and analysis: Participants will be 225 individuals with fibromyalgia recruited at Vall d'Hebron Institute of Research (Barcelona, Spain), randomly allocated to one of the three study arms: TAU vs TAU+FIBRO-On vs TAU+FIBRO-Out. A comprehensive assessment to collect functional impact, pain, fatigue, depressive-anxiety symptoms, physical function, kinesiophobia, pain catastrophism, quality of life, costs, and psychological process variables will be conducted pre-intervention, at half of the intervention (6 weeks, post-intervention (12 weeks), and at 6-month follow-up. Changes in immuno-inflammatory biomarkers (i.e. IL-6, CXCL8, IL-17A, IL-4, IL-10, and high-sensitivity C reactive protein) and Brain-Derived Neurotrophic Factor will be evaluated in 50% of the sample at pre- and post-treatment. Linear mixed-effects models using restricted maximum likelihood, mediational models and a full economic evaluation applying bootstrapping techniques, acceptability curves and sensitivity analyses will be computed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, between 18 and 65 years of age.
2. Diagnosis of fibromyalgia according to the ACR 2010/2011 criteria.
3. Understanding Spanish.

Exclusion Criteria:

1. Psychological treatment (within the last year) or current.
2. Comorbid presence of severe mental disorder (e.g. schizophrenia) or other terminal clinical conditions or scheduled treatments that may interrupt study follow-up.
3. Inability to complete the weekly sessions/modules of the programme on a regular basis.
4. Being in litigation with the health system with the aim of obtaining a permanent leave of absence.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Change from baseline values at 6 months
  The FIQR comprises three dimensions: physical dysfunction (scores from 0 to 30), overall impact (scores from 0 to 20), and intensity of the symptoms (scores from 0 to 50) is used to measure the impact generated by FM during the last week. It consists of 21 items, which are answered on a numerical rating scale of 11 points (from 0 to 10). Total scores can range from 0 to 100, with higher scores reflecting greater deterioration.

SECONDARY OUTCOMES:
Visual-analogue scale of perceived pain (VAS-Pain) | Change from baseline values at 6 months
  Patients indicate their pain during the last week on a 10 cm line. Total scores range from 0 to 10, where higher scores indicate a greater pain.
Visual-analogue scale of perceived fatigue(VAS-Fatigue) | Change from baseline values at 6 months
  Patients indicate their fatigue during the last week on a 10 cm line. Patients indicate their pain during the last week on a 10 cm line. Total scores range from 0 to 10, where higher scores indicate a greater fatigue.
Hospital Anxiety and Depression Scale (HADS) | Change from baseline values at 6 months
  HADS is used to quantify the severity of anxiety and depression symptoms. It consists of two dimensions (anxiety and depression) of 7 items each responding on a Likert scale of 4 points. Total scores of each scale (HADS-A and HADSD) range from 0 to 21, where higher scores indicate greater severity of symptoms.
Perceived Stress Scale (PSS) | Change from baseline values at 6 months
  PSS is used to evaluate the stress perceived by people during the last month. This study will use a 4 item version. The response format of this scale is 5-point Likert type. Total scores range from 0 to 16, with higher scores indicating greater perceived stress
Short Form-36 Health Survey (SF-36) | Change from baseline values at 6 months
  Physical Function of the 36-Item Short Form Survey (SF-36) was used to measure physical function.This dimension comprises a total of 10 items, which are answered on a Likert scale of 3 points. Total scores on each scale are then transformed and can range from 0 to 100, with higher scores indicate better physical function.
EuroQoL-5D (EQ-5D) | Change from baseline values at 6 months
  An instrument for assessing health-related quality of life. It consists of two parts: the first part assesses the individual's difficulties in relation to mobility, self-care, pain/discomfort and anxiety/depression; and the second part assesses the patient's current perceived health status on an analogue-visual scale from 0 to 100.
Client Service Receipt Inventory (CSRI) | Change from baseline values at 6 months
  Questionnaire for economic evaluation. The version used in this study is designed to retrospectively collect data on the use of health and social services during the previous 6 months.
Pain Catastrophising Scale (PCS) | Change from baseline values at 6 months
  PCS is used to evaluate catastrophic thoughts associated with pain. It consists of three dimensions (rumination, magnification, and helplessness) of 13 items in total, which are answered on a Likert scale of 5 points. Total scores on each scale range from 0 to 52, with higher scores indicating more catastrophic thoughts.
Psychological inflexibility in pain scale (PIPS) | Change from baseline values at 6 months
  A 12-item scale that assesses psychological inflexibility in pain patients and includes two factors: avoidance and cognitive fusion with pain. Respondents are asked to rate items on a 7-point scale that ranges from 1 (never true) to 7 (always true). Higher scores indicate greater levels of psychological inflexibility.
Tampa Scale for kinesiophobia (TSK-11) | Change from baseline values at 6 months
  TSK-11 is used to assess fear of pain and movement. It consists of 11 items, which are answered on a Likert scale of 4 points. Total scores of each scale range from 11 to 44, where higher scores indicate a greater fear of pain and movement.
The Patient Global Impression of Change (PGIC) | Change from baseline values at 6 months
  Is a measure that has been frequently used as indicators of meaningful overall change [on a 7-point Likert scale, from 1 = "Much better" to 7 = "Much worse"] in treatments for chronic pain.
Pain Specific Impression of Change (PSIC) | Change from baseline values at 6 months
  The PSIC asks about the impression of change in more specific domains than PGIC: physical and social functioning, work-related activities, mood, and pain [on a 7-point Likert scale, from 1 = "Much better" to 7 = "Much worse"].
Adverse effects of treatments | Change from baseline values at 6 months
  Ad hoc measure to check for the presence of negative effects of psychological treatments.
Socio-demographic questionnaire | Change from baseline values at 6 months
  Gender, date of birth, marital status, living arrangements, educational level and employment status.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Feliu, PhD, Principal Investigator — Universitat Autonoma de Barcelona
Locations (1):
- Hospital Vall Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferres S, Serrat M, Auer W, Royuela-Colomer E, Almirall M, Lizama-Lefno A, Nijs J, Maes M, Luciano JV, Borras X, Feliu-Soler A. Immune-inflammatory effects of the multicomponent intervention FIBROWALK in outdoor and online formats for patients with fibromyalgia. Brain Behav Immun. 2025 Mar;125:184-197. doi: 10.1016/j.bbi.2024.12.149. Epub 2024 Dec 30. PMID 39742894
- [Derived] Serrat M, Ferres S, Auer W, Almirall M, Lluch E, D'Amico F, Maes M, Lorente S, Navarrete J, Montero-Marin J, Neblett R, Nijs J, Borras X, Luciano JV, Feliu-Soler A. Effectiveness, cost-utility and physiological underpinnings of the FIBROWALK multicomponent therapy in online and outdoor format in individuals with fibromyalgia: Study protocol of a randomized, controlled trial (On&Out study). Front Physiol. 2022 Nov 10;13:1046613. doi: 10.3389/fphys.2022.1046613. eCollection 2022. PMID 36452042